CLINICAL TRIAL: NCT00094133
Title: Hypnosis for Hot Flashes in Breast Cancer Survivors
Brief Title: Hypnosis in Treating Hot Flashes in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000481365; S-WHITE-8165; NCT00324337 (obsolete NCT alias)
Record Dates: First submitted 2004-10-14; First posted 2004-10-15 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer; Cancer Survivor; Hot Flashes
Keywords: cancer survivor; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; breast cancer in situ; inflammatory breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ; Inflammatory Breast Neoplasms | interventions — Hypnosis

INTERVENTIONS:
Procedure: hot flashes attenuation
Procedure: hypnotherapy

SUMMARY:
RATIONALE: Hypnosis may be effective in decreasing hot flashes in breast cancer survivors.

PURPOSE: This randomized clinical trial is studying how well hypnosis works in treating hot flashes in breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of hypnosis in controlling hot flashes in women who are breast cancer survivors.
* Determine the extent to which hypnotizability is related to the success of the hypnotherapy intervention.

OUTLINE: This is a randomized, controlled study. Patients are stratified according to age, gender, race, and educational background. All patients complete a Hot Flash Daily Diary to record frequency and severity of hot flashes for 1 week. Patients are then randomized to 1 of 2 treatment arms.

* Arm I (hypnotherapy): Patients undergo hypnotherapy once a week for 5 weeks. Patients complete the Hot Flash-Related Daily Interference Scale, the Hospital Depression and Anxiety Sub-scale, the CES Depression Scale, and the MOS-Sleep and Sexual Function Scales in week 5 after the last hypnotherapy intervention. Patients also complete another Hot Flash Daily Diary for 1 week in week 6 and are administered the Stanford Hypnotic Clinical Scale in week 7.
* Arm II (control): Patients receive no contact for 4 weeks. Patients complete the questionnaires as in arm I in week 5. Patients also complete another Hot Flash Daily Diary for 1 week in week 6 and are administered the Stanford Hypnotic Clinical Scale in week 7.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of primary breast cancer

  * No evidence of detectable disease
* At least 14 hot flashes per week for ≥ 1 month by self-reporting
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Life expectancy > 6 months
* Menopausal status not specified
* Outpatient status
* No medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* Concurrent antihormonal agents for breast cancer (e.g., tamoxifen or raloxifene) allowed provided the patient has been on them for ≥ 1 month
* No other concurrent hormonal therapy
* No other putative therapies for hot flashes ≥ 1 month prior to study entry

  * Concurrent vitamin E allowed
* No other concurrent treatment for hot flashes
* No concurrent cytotoxic chemotherapy
* Not concurrently using hypnosis for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Hot flash control by Hot Flash Daily Diary in week 6

CONTACTS AND LOCATIONS:
Overall Officials: Gary Elkins, PhD, Principal Investigator — Scott and White Hospital & Clinic
Locations (1):
- Scott and White Cancer Institute, Temple, Texas, United States

REFERENCES:
- [Result] Elkins G, Marcus J, Stearns V, Perfect M, Rajab MH, Ruud C, Palamara L, Keith T. Randomized trial of a hypnosis intervention for treatment of hot flashes among breast cancer survivors. J Clin Oncol. 2008 Nov 1;26(31):5022-6. doi: 10.1200/JCO.2008.16.6389. Epub 2008 Sep 22. PMID 18809612